CLINICAL TRIAL: NCT00037583
Title: A Dose-Ranging Study of the Safety and Efficacy of Gemtuzumab Ozogamicin (go) Given in Combination With Cytarabine and Daunorubicin in Relapsed or Refractory Patients and in Younger de Novo Patients With Acute Myeloid Leukemia (AML)
Brief Title: Study Evaluating the Safety and Efficacy of Gemtuzumab Ozogamicin in Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Purpose: Treatment
Other Study IDs: 0903B1-206
Record Dates: First submitted 2002-05-17; First posted 2002-05-20 (Estimated); Last update posted 2009-08-21 (Estimated); Status verified 2009-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute; Myeloid; Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — Gemtuzumab

INTERVENTIONS:
Drug: Gemtuzumab Ozogamicin

SUMMARY:
The primary objectives are a) to establish the maximum tolerated dose (MTD) of gemtuzumab ozogamicin in combination with cytarabine and daunorubicin, and b) to assess the safety of gemtuzumab ozogamicin when given concurrently with cytarabine and daunorubicin.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients with relapsed or refractory AML, as well as younger de novo AML patients are eligible for the study
* Relapsed, refractory, and de novo AML patients are allowed in Phase I of this study
* Phase II will only allow enrollment of younger de novo AML

Exclusion Criteria:

* AML following an antecedent hematologic disorder (myelodysplasia or myeloproliferation) of greater than 2 months duration
* De novo patients with M3 AML
* AML secondary to exposure to chemotherapy or radiation

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

REFERENCES:
- [Derived] Hibma J, Knight B. Population Pharmacokinetic Modeling of Gemtuzumab Ozogamicin in Adult Patients with Acute Myeloid Leukemia. Clin Pharmacokinet. 2019 Mar;58(3):335-347. doi: 10.1007/s40262-018-0699-5. PMID 30062662